CLINICAL TRIAL: NCT04196166
Title: Does More Testing in Routine Preoperative Evaluation Benefit the Surgical Patient? Matched Case Control Study From a Resource-constrained Setting
Brief Title: Routine Preoperative Evaluation in Surgical Patient
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Obada Hasan, FCPS, MRCS, MSc (Epidemiology&Biostatistics), Principle Investigator, Aga Khan University
Other Study IDs: 4226-Sur-ERC-16
Record Dates: First submitted 2019-12-03; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Orthopedic Disorder
Keywords: preoperative evaluation; orthopedic surgery
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: nested from on going retrospective cohort study. Participants who had change in their surgical plan after hospitalization.
  Interventions: Other: preoperative blood tests
- Controls: nested from on going retrospective cohort study. Participants who didn't have change in their surgical plan after hospitalization.
  Interventions: Other: preoperative blood tests

INTERVENTIONS:
Other: preoperative blood tests

SUMMARY:
The "routine" pre-operative tests in healthy orthopaedic patients undergoing intermediate/ major surgery are not justified. In this study of 670 healthy orthopedic patients with 7610 preoperative tests, investigators found that surgical plan was influenced in <1% of patients. Surgeons should be sensitized to reconsider this practice particularly with limited resources.

DETAILED DESCRIPTION:
Background: Routine preoperative tests in healthy patients not only cause extra anxiety, but may delay treatment without influencing surgical plan. This has worse impact in resource-constrained settings where fee for service rather than health insurance is the usual norm. Investigators aim to determine if "routine" pre-operative tests are justified in healthy orthopedic patients.

Methods: Investigators conducted a non-commercialized, non-funded matched case control study in tertiary care university hospital and a level-1 trauma centre for healthy patients (ASA-1&2) admitted from January 2014-December 2016 for elective orthopedic intermediate and major procedures. Cases (patient who had a change in his/her surgical plan after admission) and controls were selected independently of the exposure of interest then matched randomly to cases on age, gender and procedure type. Primary exposure was the routine preoperative lab tests, as defined by the American Society of Anesthesiologist, which included 13 blood tests. Analysis was done using Principle Component Analysis and Conditional logistic regression at univariate and multivariable levels reporting matched adjusted Odds Ratios. The data will bereported in line with STROBE criteria.

.

ELIGIBILITY:
Inclusion Criteria:

* Participants irrespective of age and gender.
* ASA-1 and ASA-2 status.
* Primary elective orthopedic procedures.
* Blood lab tests done at the institution only.

Exclusion Criteria:

* Ambulatory care procedures
* Revision surgery.
* Participants admitted to other services, high care or intensive care units.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients irrespective of age and gender who were classified as ASA-1 and ASA-2 by the anesthesia team and who underwent minor, intermediate and major primary elective orthopedic procedures
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
preoperative blood tests compliance rate with institutional guidelines | 2014-2019
  compliance rate (%) with institutional and international guidelines measured by a questionnaire including whether participant was advised preoperative lab tests in compliance with the institutional guidelines or not.

SECONDARY OUTCOMES:
Cost difference in local currency | 2014-2019
  of compliant group Vs non compliant

IPD SHARING:
Plan to Share IPD: No
Not allowed by organisation